CLINICAL TRIAL: NCT07178106
Title: Investigation of the Relationship Between Peripheral and Central Metabolic Changes Caused by Fasting
Acronym: Meta-Fast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nils Opel (Other)
Collaborators: University Hospital, Bonn (Other); Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Sponsor-Investigator, Nils Opel, Prof Dr med, Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-3502_1-BO
Record Dates: First submitted 2025-01-17; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Fasting; MR Spectroscopy; fMRI; Metabolism; Autophagy; Immune response
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group/ Arm (Experimental): Healthy participants
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Participants undergo the standardised Wilhelmi-Buchinger fasting intervention, which consists of two days of preparation with a dietary energy supply of <1000 kcal, three days of fasting with a dietary energy supply of 300-500 kcal with tea, broth, fruit and vegetable juices, and two days of recovery.
  Other Names: Wilhelmi-Buchinger-fasting

SUMMARY:
Fasting has become an increasingly popular intervention for improving both physical and mental health. This study aims to explore the biological mechanisms underlying the positive effects of low caloric fasting (Wilhelmi-Buchinger-fasting). Specifically, we focus on the metabolic transition from glucose to fat utilization and its effects on systemic and brain metabolism. By examining the relationship between peripheral metabolic changes and brain metabolism, this research aims to uncover how these shifts influence brain metabolism and behaviour.

DETAILED DESCRIPTION:
Therapeutic fasting, specifically Buchinger fasting, is a widely recognized method in integrative medicine. It is frequently used to treat a variety of chronic diseases, including inflammatory and metabolic disorders. In addition to its benefits for physical health, fasting is increasingly recognized for its potential to improve mental health.

Research has shown that fasting can induce significant biological effects, including the metabolic switch, which involves the transition from glucose to fat as the primary energy source. This shift typically occurs around day two of the fasting period and has important implications for peripheral metabolism. However, little is known about how these peripheral metabolic changes are linked to brain metabolism and how this connection might affect brain network function and, ultimately, psychological and cognitive processes.

Recent studies have shown that fasting influences both peripheral metabolism and brain function, with potential benefits for mental health. The precise mechanisms and timing of these changes remain unclear. The current study will focus on understanding (i) how peripheral metabolic changes during fasting relate to central metabolic changes in the brain, (ii) how these changes affect brain network function over time, and (iii) the connection between these metabolic and functional brain changes with psychological and cognitive alterations during fasting.

This study will use detailed metabolic profiling and neuroimaging techniques, alongside psychological assessments, to explore these complex interactions in healthy, fasting individuals, providing a foundation for further research into its potential as an intervention for mental health disorders.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight at study inclusion (BMI 18.5-25)
* Generally good physical condition without serious previous illnesses
* For female participants, only participants taking hormonal contraception are included

Exclusion Criteria:

* MRI contraindication: cardiac pacemakers, hearing aids, neurostimulation, insulin pumps, other potentially ferromagnetic implants, screws, clips, prostheses, metal splinters, etc., pregnancy, claustrophobia, extensive tattoos, medication that impairs thermoregulation
* Comorbidity: neurological or psychiatric conditions, cognitive impairments, chronic somatic disorders
* Intake of more than 40g of pure alcohol (for men) or more than 20g of pure alcohol (for women), smoking, regular drug use
* Pregnancy or nursing
* Current or within the past five years eating disorder, vegan diet or fasting within the past six months
* Regular medication intake

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
MR spectroscopy | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  metabolites between 0-4 ppm in regions including the posterior cingulate cortex (PCC), medial cingulate cortex (MCC), and anterior insula

SECONDARY OUTCOMES:
Structural MR imaging | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  cortical thickness, grey matter volume
Functional MRI | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  resting state functional connectivity
Exploratory Proteomics of Autophagy Processes II | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  protein levels and protein phosphorylation by targeted and untargeted mass spectrometry-based proteomics and phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells)
Exploratory Proteomics of Autophagy Processes I | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  protein levels of autophagy biomarkers (e.g. LC3II & p62) of isolated PBMCs (peripheral blood mononuclear cells) by Western Blotting
Neuropsychology: Verbal Fluency | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  MWT-B, Regensburg Word Fluency Test. A composite score for verbal fluency will be derived from the Regensburg Word Fluency Test and the MWT-B. First, raw scores for each test will be converted to standardized scores (e.g., z-scores). If needed, scores will be adjusted so that higher values consistently represent better performance. The standardized scores will then be averaged to create a single composite measure of verbal fluency.
Neuropsychology: Memory | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  VLMT-A, block span. A composite memory score will be computed from the VLM-T and Block Span test. Raw scores from each test will be standardized (e.g., into z-scores). These z-scores will then be averaged to yield a single measure of memory performance, reflecting both verbal and visuospatial working memory components.
Neuropsychology: Processing speed | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Number Symbol Test, Letter-Number-Symbol Test, TMT-A. A composite score for processing speed will be derived from the Number Symbol Test, Letter-Number Symbol Test, and TMT-A. First, raw scores from each test will be normalized (e.g., converted into z-scores), taking into account that lower completion times on the TMT-A indicate better performance. The normalized scores will then be combined-after adjusting the direction of scores if necessary-by calculating their average to yield a single, unified measure of processing speed.
Neuropsychology: Attention | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  TMT-B, D2-Test. A composite attention score will be created using the D2-Test and TMT-B. Raw scores from both tests will be standardized (e.g., as z-scores). For tests such as the TMT-B, if necessary, the scores will be adjusted (e.g., reverse-coded) so that higher values indicate better attention performance. The resulting standardized scores will be averaged to form a unified attention measure.
Sleep | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Pittsburgh Sleep Quality Index (PSQI). The 19 self-rated questions of the PSQI are grouped into 7 components. Each component is scored from 0 to 3 points. The scores of the 7 components are then summed to yield a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Depression | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Beck's depression inventory (BDI-II). The questionnaire consists of 21 questions. Each question is scored on a 4-point scale ranging from no impairment (0) to severe impairment (3). The maximum score is 63.
Anxiety | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  State-Anxiety Inventory (STAI-S). For the STAI-S assessment, specific items (1, 2, 5, 8, 10, 11, 15, 16, 19, and 20) were reverse-coded because they represent aspects of anxiety expressed in a negative direction. After recoding, responses for all STAI-S items were summed to obtain the final test score for state anxiety.
Anhedonia | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Snaith-Hamilton-Pleasure-Scale (SHAPS). For scoring, each non-affirmative response ("does not apply" or "does not apply at all") is assigned 1 point, while each affirmative response is assigned 0 points. The points are summed across all items, resulting in a total score ranging from 0 to 14, with higher scores indicating a greater degree of anhedonia.
Life quality | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Positive Mental Health Scale. 9 items rated on a 4-point Likert scale ranging from 0 ("do not agree") to 3 ("completely agree"). A total score is computed by summing the responses to all items, with higher scores indicating greater positive mental health.
Numeric Analog Scales | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Assessing mood on 0-10 points and sleep duration on 0-13 points scale
Metabolic processes | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Targeted and quantitative analysis by mass spectrometry of change in metabolites of plasma
Fatigue | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Fatigue Assessment Scale (FAS), 10-item self-assessment scale. For scoring, responses to items 1-3 and 5-9 are rated on a scale from 1 to 5, while items 4 and 10 are reverse-coded (scored from 5 to 1). The scores for all items are then summed to produce the total FAS score.
Lipid profiling | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Targeted and quantitative analysis by mass spectrometry of change in plasma lipids
Transcription expression patterns | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Change of the gene expression profile by RNA sequencing of isolated PBMCs (peripheral blood mononuclear cells)
Proteome/phosphoproteome/ubiquitinome patterns | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  proteome expression patterns through blood (PBMCs and Plasma) based proteome, phosphoproteome, and ubiquitinome analysis
Exosomal protein patterns | Outcome measures are assessed as changes from baseline over 3 fasting days, with follow-up on day 4 during refeeding, during a one-week on-site visit per participant, within an overall study period of 2 months
  Evaluate exosomal protein content through blood based metabolome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sharmili Edwin Thanarajah, PD Dr med, Principal Investigator — Goethe University; Nils Gassen, Prof Dr, Principal Investigator — University Hospital, Bonn
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Jena, Jena, Thuringia, Germany